CLINICAL TRIAL: NCT03612973
Title: Assessment of Changes in Liver Fibrosis and Stiffness, Lipid Profile and Insulin Resistance in Patients With Chronic Hepatitis C Viral Infection Who Received Direct Acting Antiviral Therapy
Brief Title: Changes in Liver Fibrosis, Lipid Profile and Insulin Resistance in HCV Patients Who Received Antiviral Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa hanafy, principal investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: assuit 1234
Record Dates: First submitted 2018-07-23; First posted 2018-08-02 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Chronic Hepatitis c
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Intervention Model Description: both study groups will be investigated at same time
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- non cirrhotic HCV patients (Active Comparator): * complete blood picture
  * Liver and renal function tests
  * Prothrombin time and concentration
  * HCV quantitative polymerase chain reaction
  * Hepatitis B surface Ag
  * lipid profile
  * fasting blood glucose level
  * fasting insulin level
  * homeostasis model for the assessment of insulin resistance (HOMA-IR)
  * fibrosis (FIB- 4) index
  * Aspartate aminotransferase (AST)/platelet ratio index (APRI)
  * Abdominal ultrasound to assess liver and spleen
  * Fibroscan/transient elastography to grade hepatic fibrosis all these investigations will be done before and after receiving direct acting antiviral therapy (sofosbuvir 400 mg once daily + daclatasvir 60 mg once daily) for 12 weeks
  Interventions: Diagnostic Test: lipid profile; Diagnostic Test: fasting insulin; Diagnostic Test: fibro scan
- cirrhotic HCV patients (Active Comparator): * complete blood picture
  * Liver and renal function tests
  * Prothrombin time and concentration
  * HCV quantitative polymerase chain reaction
  * Hepatitis B surface Ag
  * lipid profile
  * fasting blood glucose level
  * fasting insulin level
  * homeostasis model for the assessment of insulin resistance (HOMA-IR)
  * Fibrosis (FIB- 4) index
  * Aspartate aminotransferase (AST)/platelet ratio index (APRI)
  * Abdominal ultrasound to assess liver and spleen
  * Fibroscan/transient elastography to grade hepatic fibrosis all these investigations will be done before and after receiving direct acting antiviral therapy (sofosbuvir 400 mg once daily + daclatasvir 60 mg once daily) for 12 weeks
  Interventions: Diagnostic Test: lipid profile; Diagnostic Test: fasting insulin; Diagnostic Test: fibro scan

INTERVENTIONS:
Diagnostic Test: lipid profile — Serum samples will be withdrawn after fasting 12 hours then performed on Siemens Dimension Max: Total cholesterol and triglyceride concentrations will be estimated using enzymatic methods ( Roche Diagnostics, Mannheim, Germany). High density lipoprotein cholesterol will be determined after precipitation with phosphotungstic acid/magnesium chloride. Low density lipoprotein(LDL) cholesterol will be measured directly with a commercially available direct LDL-C assay (LDL-C Plus assay; Roche Diagnostics)
Diagnostic Test: fasting insulin — serum samples used for doing the test by ELISA after fasting for 8 h
Diagnostic Test: fibro scan — liver stiffness by fibro scan before and after treatment

SUMMARY:
Hepatitis C virus (HCV) is one of the major globally cause of death and morbidity.Chronic hepatitis C is the leading cause of end-stage liver disease, hepatocellular carcinoma and liver-related death in Egypt.It could be considered a special type of metabolic diseases involving insulin resistance (IR) which accelerates fibrosis and modulation of lipid-cholesterol biosynthesis with increased risk for ischemic heart diseases.It could be considered a special type of metabolic diseases involving insulin resistance (IR) which accelerates fibrosis and modulation of lipid-cholesterol biosynthesis with increased risk for ischemic heart diseases .Increased prevalence of IR and type 2 diabetes mellitus extensively reported in HCV infections

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) is one of the major globally cause of death and morbidity and recent estimates showed increase in its prevalence over the last decade to > 185 million infections worldwide. Prevalence HCV infection in Egypt is the highest in the world.Chronic viral hepatitis infection increases liver fibrosis and stiffness and is an important cause of liver cirrhosis. Chronic hepatitis C is the leading cause of end-stage liver disease, hepatocellular carcinoma and liver-related death in Egypt.It could be considered a special type of metabolic diseases involving insulin resistance (IR) which accelerates fibrosis and modulation of lipid-cholesterol biosynthesis with increased risk for ischemic heart diseases .Increased prevalence of IR and type 2 diabetes mellitus extensively reported in HCV infections.Interferon (INF) based therapy was used in chronic HCV patient and investigators reported that it's effective in eradicating HCV RNA and improving liver fibrosis. However, It's associated with several side effects.Novel direct antiviral agents (DAA) for chronic hepatitis C have entered clinical practice. This therapeutics has minimal side effects and achieves sustained virological response (SVR) rates of above 90% of patients and they are shorter and simpler regimens.Liver fibrosis severity assessment is important when staging chronic HCV and it reflects impact of serological viral eradication on hepatic damage and fibrosis. Although liver biopsy is the gold standard procedure for fibrosis assessment, but non-invasive new approaches have been strongly recommended for evaluation of fibrosis, mainly in HCV. They have no complications and have good diagnostic accuracy. One of the most used non-invasive mechanical methods based on ultrasound is transient elastography (Fibro Scan). Although association of baseline metabolic characteristics with treatment outcome has not been fully assessed for DAAs, this group was reported to result in improved rates of SVR and to reduce the predictive ability of these factors except for the baseline low density lipoprotein. The highest prevalence of HCV was reported in Egypt, where genotype 4 is responsible for 91% of infections and DAAs represented main line of treatment in most centers.Although the changes in lipid metabolism after treatment with DAAs were reported for other genotypes. It was not fully studied in genotype 4 infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 ys.
* Disease status: patients with chronic hepatitis C infection, based on the presence of anti-HCV and detectable serum HCV-RNA for 6 months or more who had different grades of fibrosis (F) as estimated by fibroscan
* Treatment: treatment naïve patients who will receive direct acting antiviral drugs (Sofosbuvir and Daclatasvir ± ribavirin) for 12 weeks
* Negative hepatitis B virus surface Ag and HIV antibodies
* No history of hepatocellular carcinoma or development of hepatocellular carcinoma during the treatment period
* No other causes of chronic liver disease (alcohol consumption more than 80 g/day, hepatotoxic drugs, autoimmune hepatitis, primary biliary cholangitis, hemochromatosis and Wilson's disease).

Exclusion Criteria:

* Diabetic patients.
* Patients using lipid lowering agents.
* HCV co-infection with hepatitis B virus(HBV) or human immunodeficiency virus(HIV)
* Presence of other causes of chronic liver disease (alcohol consumption more than 80 g/day, hepatotoxic drugs, autoimmune hepatitis, primary biliary cholangitis, hemochromatosis and Wilson's disease).
* Patients with hepatocellular carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in liver fibrosis in HCV patients after receiving direct acting antiviral therapy | 1 year
  by using non-invasive measures (fibro scan) before and after end of treatment (12 weeks0

SECONDARY OUTCOMES:
Effect of HCV treatment by direct acting antiviral therapy on lipid profile of chronic HCV patients | 1 year
  changes in values of total cholesterol, triglycerides, LDL and HDL at the baseline and end of treatment (12 weeks)
Changes and degree of improvement in insulin resistance in HCV patients after receiving direct acting antiviral therapy | 1 year
  measuring fasting insulin and glucose level with calculation of homeostasis model for the assessment of insulin resistance at the baseline and end of treatment (12 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospital, Asyut, Egypt